CLINICAL TRIAL: NCT02882451
Title: Impact of Pinaverium Bromide on Bile Duct and Pancreatic Duct Cannulation During Endoscopic Retrograde Cholangiopancreatography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Head of Digestive Endoscopy Center, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERCP-02
Record Dates: First submitted 2016-07-22; First posted 2016-08-29 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Bile Duct Diseases
Keywords: bile duct; endoscopic retrograde cholangiopancreatography; pinaverium bromide
MeSH Terms: conditions — Bile Duct Diseases | interventions — pinaverium; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pinaverium bromide (Experimental): take 50 mg pinaverium bromide three times a day 1 days before and then 100 mg 1 hour before the examination orally
  Interventions: Dietary Supplement: pinaverium bromide
- Vitamin C (Placebo Comparator): take 50 mg Vitamin C three times a day 1 days before and then 100 mg 1 hour before the examination orally
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: pinaverium bromide
  Arms: pinaverium bromide
Dietary Supplement: Vitamin C
  Arms: Vitamin C

SUMMARY:
Pinaverium bromide can be used to treat symptoms related to irritable bowel syndrome (IBS) and functional disorders of the biliary tract. In this study, pinaverium bromide was compared with Vitamin C for the facilitation of bile duct and pancreatic duct cannulation in patients. The primary outcome was successful deep bile duct cannulation and pancreatic duct canulation. The second outcome was the major papillary orifice,bile juice flow from the papilla, time to achieve deep bile duct cannulation, fluoroscopy time for deep bile duct cannulation,the appearance of the major and minor papillary orifice, pancreatic juice flow from the papilla, time to achieve deep pancreatic duct cannulation, and fluoroscopy time for deep pancreatic duct cannulation in the pinaverium bromide group versus Vitamin C group.

ELIGIBILITY:
Inclusion Criteria:

1. those with intact native papilla,
2. who underwent endoscopic retrograde choledochopancreatography for bile duct,
3. age≥18 years, ≤80years, and
4. agreement to participate in the study.

Exclusion Criteria:

1. a previous sphincterotomy,
2. previous attempted or unsuccessful endoscopic retrograde choledochopancreatography with papillary manipulation,
3. indwelling biliary or pancreatic stent(s),
4. active acute pancreatitis,
5. active acute pancreatitis
6. altered/postsurgical anatomy,
7. history of gastroparesis,
8. endoscopic retrograde choledochopancreatography for sphincter of Oddi's sphincter(SO) manometry,
9. known tumor of the major duodenal papilla, and
10. patients with any medication probably affecting SO motility

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
cannulation time for deep bile duct cannulation and pancreatic duct cannulation | 2 days

SECONDARY OUTCOMES:
bile juice flow from the major papilla and pancreatic juice flow from the major papilla | 2 days
appearance of the major papillary orifice | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China